CLINICAL TRIAL: NCT04241445
Title: Tracking General Movements: An Observing-the-Observer Approach to Enhance Clinical Reasoning
Brief Title: Tracking General Movements
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 30-261 ex 17/18
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Clinical Reasoning; Cerebral Palsy; General Movement Assessment
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- novice observers: who have practiced GMA sporadically (def.: < = 2 GMA/week for < = 2 years), have limited experience, and do not use GMA in clinical settings
- GMA experts: GMA tutors and individuals who have applied GMA regularly (def.: > 2 GMA/week for > 2 years)

SUMMARY:
Background: General movements (GMs) are endogenously generated movements of the entire body observable from the 9th week postmenstrual age to at least 20 weeks postterm age. The assessment of GMs, the GMA, is a method to differentiate between spontaneous normal vs. abnormal motor patterns based on visual Gestalt perception, and has proven to be a reliable tool to evaluate the integrity of the nervous system in early infancy. Trained GMA observers achieve an excellent inter-observer agreement, but this accuracy is known to decline when GMA is applied infrequently. Although specific changes in the quality of GMs are highly predictive for atypical neurodevelopmental trajectories, one pattern of GMs, the poor-repertoire, is still of low predictive power.

Objectives: Tracking GMA observers' intrinsic and unconsciously applied analytic strategies may unravel hitherto unknown characteristics of GMs and Gestalt perception in clinical reasoning. We specifically aim to: detect parameters during the writhing movements period which differentiate normalising and deteriorating developmental trajectories (Aim 1); evaluate different strategies/modalities of expert guidance for clinical reasoning and develop novel didactical approaches for remote GMA training (remote visual and verbal guidance; Aim 2); create a database to provide expert-guided tutorials for remote clinical training, observer re-calibration, and self-evaluation for certified observers (Aim 3).

DETAILED DESCRIPTION:
Approach / methods: Based on our expertise in GMA and eye tracking, and a successful proof of principle (pilot experiment), we will conduct a series of experiments: GMA experts' eye movement patterns during clinical reasoning will be assessed to better understand the diagnostic category of poor-repertoire GMs (Experiment 1); benefits and potential difficulties of different modes of "seeing through the eyes of an expert"-approaches for GMA-training will be explored (Experiment 2); we shall evaluate enhancement of clinical reasoning as a result of intensive remote GMA training (Experiment 3).

Level of originality / innovation: "Tracking general movements" will (1) contribute to better understand poor-repertoire GMs adding to the clinical necessity to closely follow infants in need for continuous or close-meshed clinical surveillance; (2) define the benefits of different modes/modalities of expert guidance for GMA, which will form the basis for innovative remote clinical GMA training; and (3) create a globally accessible database for remote clinical GMA refreshment-training and re-calibration.

ELIGIBILITY:
Inclusion Criteria:

Observers have to provide written informed consent to the study protocol, data analysis and data storage guidelines, as well as the publication of study results.

Observers have to complete the experimental data acquisition. Apart from their lack of GMA training, naïve observers have to be of the same gender, of comparable age and educational level as GMA-trained observers.

Novice observers and GMA experts have to be certified for GMA. Observers must have normal or corrected-to-normal vision (only individuals wearing soft contact lenses can be included in the eye tracking experiments).

Exclusion Criteria:

Observers did not adhere to the study protocol, data analysis, data storage guidelines, or the publication of study results.

Observers did not complete the experimental data acquisition. Observers have uncorrected visual impairments or visual impairments corrected with glasses/hard contact lenses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the proposed experiments, observers will be divided into three groups. One group will consist of (a) naïve observers, that is, individuals who are not familiar with GMs, have not received any GMA training and are not medically educated. The two other groups will consist of (b) GMA-trained and certified observers: (b1) novice observers who have practiced GMA sporadically (def.: <= 2 GMA/week for <= 2 years) and have only little experience; and (b2) GMA experts, i.e. GMA tutors and individuals who have applied GMA regularly (def.: > 2 GMA/week for > 2 years).
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Spotlight on the very early motor repertoire: writhing general movements (WMs); GMA experts only | 1st - 16th month
  Detect parameters during the WMs period which differentiate normalising and deteriorating GM traits by experts
Expert-guided clinical reasoning - "seeing through the eyes of an expert" | 21st - 32rd month
  Develop and provide expert-guided video recordings to complement GMA trainings with three modes of visual expert guidance (i: verbal; ii: visual; iii: verbal+visual) to enhance clinical reasoning in novice observers
Implementation of a database and intensive remote GMA training | 17th - 48th month
  Create the prototype of a password-protected database for clinical GMA training. The database will cover three distinct aspects of GMA training: (i) expert-guided remote training, (ii) re-calibration, and (iii) self-evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- MUGraz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No